CLINICAL TRIAL: NCT05134168
Title: Ligation of Intersphincteric Fistula Tract (LIFT) With or Without Injection of Bone Marrow Mononuclear Cells in Treatment of Trans-sphincteric Anal Fistula; a Randomized Controlled Trial
Brief Title: LIFT With or Without Injection of BM-MNCs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Associate professor of surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mansoura2022LIFT
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIFT (Active Comparator): Patients underwent LIFT proecdure
  Interventions: Procedure: LIFT
- LIFT+bone marrow mononuclear cell injection (Active Comparator): Patients underwent LIFT with bone marrow mononuclear cell injection
  Interventions: Procedure: bone marrow mononuclear cell injection; Procedure: LIFT

INTERVENTIONS:
Procedure: bone marrow mononuclear cell injection — bone marrow mononuclear cells were injected in the intersphincteric space and around the internal opening after ligation and division of the tract
  Arms: LIFT+bone marrow mononuclear cell injection
Procedure: LIFT — The fistula tract is ligated in the intersphincteric space

SUMMARY:
To improve the outcome of LIFT, some authors used a combined approach of LIFT. Pooled analysis of seven studies including 192 patients revealed a success rate of 83.5 % after combined LIFT approach. The use of bone marrow aspirate concentrate (BMAC) in surgery is not entirely new as it has been widely used in the treatment of bone defects, mandibular reconstruction, maxillary sinus augmentation and in critical limb ischemia.

A previous study concluded that the use of BMAC to augment external anal sphincter repair strengthens wound healing by transferring cells responsible for healing directly to the site of repair. The current study aimed to assess the outcome of local injection of bone marrow mononuclear cells (BM-MNCs) in conjunction with LIFT as compared to LIFT alone in regards to healing rate, time to healing, and ultimate success rate.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of either gender presented with cryptoglandular trans-sphincteric anal fistula

Exclusion Criteria:

* Patients with secondary anal fistula
* Immunocompromised patients
* Patients with previous pelvic radiotherapy
* Pregnant women
* Patients with ASA (American society of anesthesiologists) III or higher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with complete healing of anal fistula as assessed by clinical examination | 6 months
  Healing is defined as complete epithelization of the anal wound with absence of fistula tract

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided